CLINICAL TRIAL: NCT03791463
Title: A Phase I, Single Centre, Randomized, Open-Label, Three-Period Crossover Study to Investigate the Effect of Food on Pharmacokinetics of Salvianolic Acid A in Healthy Subjects
Brief Title: Effect of Food on Pharmacokinetics of Salvianolic Acid A in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Cui Yimin, Director of pharmacy, M.D & Ph.D, Peking University First Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAA002
Record Dates: First submitted 2018-12-20; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — salvianolic acid A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- After meal (Experimental): Each subject will receive a single oral dose of 90 mg salvianolic acid A. Each dose will be administered after consumption of a low calorie, low-fat breakfast (within 30 minutes after starting food intake).
  Interventions: Drug: salvianolic acid A
- Fasting (Experimental): Each subject will receive a single oral dose of 90 mg salvianolic acid A. Each dose will be administered at the end of a 10-hour fast.
  Interventions: Drug: salvianolic acid A

INTERVENTIONS:
Drug: salvianolic acid A — Following an overnight fast of at least 10 hours, a single dose of 90 mg salvianolic acid A will be administered on 2 separate occasions (fasting and after meal) in a randomized crossover fashion with different food restrictions.

SUMMARY:
This study is an open-label, randomized, cross-over design with two single-dose treatment periods and a washout of at least 3~5 days in between each treatment visit. The study period consists of 3 visits to the study centre: Visit 1 (enrolment), Visit 2 (first single-dose treatment), Visit 3 (second single-dose treatment).

Target subject population is healthy subjects aged 18-45 years. Following an overnight fast of at least 10 hours, a single dose of 90mg salvianolic acid A will be administered on 3 separate occasions (fasting, before meal, and after meal) in a randomized crossover fashion with different food restrictions.

ELIGIBILITY:
Inclusion Criteria:

1. healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥19.0 and ≤25.0 kg/m2 at screening
2. The subject is able to communicate well with the investigator and is able to complete the trial in accordance with the protocol.

Exclusion Criteria:

1. Planned for pregnancy or pregnant within 6 months after enrollment throughout the trial.
2. Subject has any clinically significant abnormal finding on the physical exam at screening or admission.
3. Subject has a positive screening test for alcohol or drugs of abuse at screening or admission.
4. Allergic to the body.
5. Participated in any clinical trial within 3 months prior to the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
The Effect of Food Timing (Fasting and After Meal) on Pharmacokinetics of salvianolic acid A in Healthy Subject | Hour 24
  To assess the effect of food by evaluating the area under the plasma concentration versus time curve, from time zero to the time of the last quantifiable analyte concentration (AUC(0-last))

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaocong Pang, Beijing, China